CLINICAL TRIAL: NCT02703311
Title: REPAIR - transcatheteR rEPair of mitrAl Insufficiency With caRdioband System
Acronym: REPAIR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Edwards acquired Valtech Cardio Ltd in 2017 and opted to replace this study with NCT03600688.11 patients were enrolled in REPAIR and follow-up is complete.
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CB1-3
Record Dates: First submitted 2016-02-22; First posted 2016-03-09 (Estimated); Results first posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-10

CONDITIONS: Mitral Valve Insufficiency; Cardiac Valve Annuloplasty; Mitral Valve Annuloplasty; Cardiovascular Diseases; Heart Diseases; Heart Valve Diseases; Mitral Regurgitation
Keywords: Valtech Cardio; Cardioband; Mitral Valve
MeSH Terms: conditions — Mitral Valve Insufficiency; Cardiovascular Diseases; Heart Diseases; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardioband procedure (Other): Mitral valve repair with Cardioband implanted via transcatheter procedure under transesophageal echocardiography (TEE) and fluoroscopy guidance
  Interventions: Device: Cardioband

INTERVENTIONS:
Device: Cardioband — Mitral valve repair with Cardioband implanted via transcatheter procedure under transesophageal echocardiography (TEE) and fluoroscopy guidance

SUMMARY:
The Cardioband Transcatheter System (Cardioband) is indicated for the treatment of secondary (functional) mitral regurgitation (FMR). The Cardioband is a transcatheter system, deployed on the beating heart through a transseptal approach. The Cardioband is deployed along the posterior annulus of the mitral valve (MV) and is adjusted under trans-esophageal guidance on the beating heart. A CE mark study with 30 subjects has been completed and documented reduction of severity of mitral regurgitation (MR) and improvement in 6- minute walk test in subjects with moderate to severe MR.

Study objectives are to test the efficacy of the Cardioband in improving MR and heart failure symptoms in patients with symptomatic (New York Heart Association (NYHA) Class III-IVa), severe MR in the post-marketing setting, And to evaluate the safety of the Cardioband system in the post-marketing setting.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Severe (3+ to 4+) secondary Mitral Regurgitation
3. Symptomatic heart failure (NYHA Class III-IVa) despite guideline directed medical therapy including CRT if indicated
4. The Local Site Heart Team concur that surgery will not be offered as a treatment option and that medical therapy is the intended therapy.
5. Transfemoral access and transseptal deployment of the Cardioband is determined to be feasible
6. Subject is willing and able to provide informed consent and follow protocol

Exclusion Criteria:

1. EF < 20%
2. LVEDD ≥ 70 mm
3. Heavily calcified annulus or leaflets
4. Significant CAD requiring revascularization
5. Active bacterial endocarditis
6. Any percutaneous coronary, carotid, endovascular intervention or carotid surgery within 30 days or any coronary or endovascular surgery within 3 months
7. Renal insufficiency requiring dialysis
8. Life expectancy of less than twelve months
9. Subject is participating in concomitant research studies of investigational products that have not reached their primary endpoint
10. Pulmonary hypertension ≥ 70mmHg at rest
11. Mitral valve anatomy which may preclude proper device treatment
12. Right-sided congestive heart failure with echocardiographic evidence of severe right ventricular dysfunction and/or severe tricuspid regurgitation
13. Severe liver disease
14. Patient is pregnant or lactating
15. Hypersensitivity to Nickel or Chromium
16. Clinically significant bleeding diathesis or coagulopathy
17. History of mitral valve repair
18. TIA or CVA within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- Bichat hospital, Paris, France
- Germany (8):
  - Bad Nauheim, Kerckhoff-Klinik, Bad Nauheim
  - Bonn University, Bonn
  - Koln, Universitätsklinikum, Cologne
  - Universitätsklinikum Gießen und Marburg, Giessen
  - University Hospital Halle (Saale), Halle
  - Asklepios Klinik, St. Georg, Hamburg
  - Universitäres Herzzentrum Hamburg GmbH, Hamburg
  - Universitatsmedizin Mainz, Mainz
- Hospital san raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Cardioband: Patients who were enrolled and had the Cardioband procedure attempted
Period: Overall Study
Arm/Group | Cardioband
Started | 11
Implanted | 11
30 Day Follow-Up Completed | 9
Completed (Completed Study (2 years)) | 3
Not Completed | 8
Not completed — Death | 5
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Cardioband
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.9 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
EuroScore II [Mean (Standard Deviation); unit: units on a scale] — The European System for Cardiac Operative Risk Evaluation (EuroSCORE) II is a risk model which allows the calculation of the risk of death after a heart operation.
  EuroScore II risk levels are as follows:
  Low risk: <8
  Moderate risk: 8-10
  High risk: >10
  units on a scale | 7.1 (5.3)
NYHA Functional Class III or IV [Count of Participants; unit: Participants] — NYHA Classification - The stages of heart failure:
  Class I - No symptoms and no limitation in ordinary physical activity.
  Class II - Mild symptoms and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity. Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest.
  Participants | 11
Ischemic Etiology of Regurgitation [Count of Participants; unit: Participants] | 4
Dilated Cardiomyopathy [Count of Participants; unit: Participants] | 5
Previous Coronary Artery Bypass Graft [Count of Participants; unit: Participants] | 4
Chronic Renal Disease [Count of Participants; unit: Participants] | 8
Paroxysmal, Persistent, Chronic Atrial Flutter/Fibrillation [Count of Participants; unit: Participants] | 10

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Severity of MR at 30 Days of at Least One Category on a 0-4 Scale.
Description: Percentage of Patients with Reduction in MR Severity of at least one grade at 30 days compared to baseline
Time Frame: 30 days
Population: Intra-subject comparison of patients with paired data at baseline and 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cardioband
Number analyzed (Participants) | 7
Participants | 4

2. Secondary Outcome: Change in Distance Walked on 6 Minute Walk Test
Description: Median distance in meters walked during 6 Minute Walk Test (6MWT) at 6 months compared to baseline
Time Frame: 6 months over Baseline
Population: Intra-subject comparison of patients with paired data at baseline and 6 months
Measure: Median (Standard Deviation); unit: Meters
Arm/Group | Cardioband
Number analyzed (Participants) | 6
Meters | 30.7 (60.4)

3. Secondary Outcome: Change in Mitral Regurgitation Severity
Description: Mitral Regurgitation at 6, 12, and 24 months compared to baseline
Time Frame: 6, 12, and 24 months over baseline
Population: This planned endpoint of change mitral regurgitation severity in was unable to be analyzed due to the small sample size that was achieved in this study. Data available at each time point were reported as number of patients with MR grades None/Trace, Mild, Moderate, Severe.
Measure: Count of Participants; unit: Participants
Arm/Group | Cardioband
Number analyzed (Participants) | 9
Participants
  Baseline: None/Trace | 0
  Baseline: Mild | 2
  Baseline: Moderate | 4
  Baseline: Severe | 3
  6 Months: number analyzed (Participants) | 5
  6 Months: None/Trace | 1
  6 Months: Mild | 3
  6 Months: Moderate | 1
  6 Months: Severe | 0
  12 Months: number analyzed (Participants) | 3
  12 Months: None/Trace | 0
  12 Months: Mild | 3
  12 Months: Moderate | 0
  12 Months: Severe | 0
  24 Months: number analyzed (Participants) | 0

4. Other Pre Specified Outcome: Change in Distance Walked on 6 Minute Walk Test
Description: Median distance in meters walked during 6 Minute Walk Test (6MWT) at 12 and 24 months compared to baseline
Time Frame: 12, and 24 months over baseline
Population: This planned endpoint was unable to be analyzed due to the small sample size that was achieved in this study
Arm/Group | Cardioband
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Change in Quality of Life (QoL) as Measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: Median KCCQ Score. The KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Scores range from 0-100, in which higher scores reflect better health status.
Time Frame: 6, 12, and 24 months over baseline
Population: This planned endpoint was unable to be analyzed due to the small sample size that was achieved in this study
Arm/Group | Cardioband
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Change in New York Heart Association (NYHA) Class
Description: NYHA Class at 6, 12, and 24 months compared to baseline
Time Frame: 6, 12, and 24 months over baseline
Population: This planned endpoint was unable to be analyzed due to the small sample size that was achieved in this study
Arm/Group | Cardioband
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Change in Left Ventricular End Diastolic Volume (LVEDV)
Description: Median LVEDV data, as measured by TTE at 6, 12, and 24 months compared to baseline
Time Frame: 6, 12, and 24 months over baseline
Population: This planned endpoint was unable to be analyzed due to the small sample size that was achieved in this study
Arm/Group | Cardioband
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Change in Left Ventricular End Systolic Volume (LVESV)
Description: Median LVESV data, as measured by TTE at 6, 12, and 24 months compared to baseline
Time Frame: 6, 12, and 24 months over baselines
Population: This planned endpoint was unable to be analyzed due to the small sample size that was achieved in this study
Arm/Group | Cardioband
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Number of Participants With Device Success
Description: Device success is defined as deployment of the Cardioband, with MR reduction at hospital discharge.
Time Frame: Discharge
Population: The outcome is reported for subjects where data is available. Subjects with missing data are excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cardioband
Number analyzed (Participants) | 8
Participants | 7

10. Other Pre Specified Outcome: Number of Participants With Patient Success
Description: Individual patient success (measured at 6 months and 1 year) defined as device success and the following:
  * Discharged from index hospitalization
  * NYHA class improvement by at least 1 level from baseline
Time Frame: 6 and 12 months
Population: The outcome is reported for subjects where data is available. Subjects with missing data are excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cardioband
Number analyzed (Participants) | 5
Participants
  6 Months | 3
  12 Months: number analyzed (Participants) | 4
  12 Months | 3

11. Other Pre Specified Outcome: Number of Days Alive and Out of Hospital
Description: Days alive and out of hospital due to major cardiovascular events at 1 year
Time Frame: 12 months
Population: This planned endpoint was unable to be analyzed due to the small sample size that was achieved in this study
Arm/Group | Cardioband
Number analyzed (Participants) | 0

12. Other Pre Specified Outcome: Freedom From All-cause Mortality and Major Adverse Events (AE)
Description: Freedom from all-cause mortality and major AE is defined as disabling stroke, myocardial infarction (MI) (peri-procedural or spontaneous), renal failure requiring dialysis, life-threatening bleeding, cardiac tamponade and device related cardiac surgical intervention at 30 days from the implant procedure or hospital discharge, whichever is later.
Time Frame: 30 days from implant procedure or hospital discharge, whichever is later.
Measure: Count of Participants; unit: Participants
Arm/Group | Cardioband
Number analyzed (Participants) | 11
Participants | 10

13. Other Pre Specified Outcome: Need for Urgent/Emergent Surgical Intervention
Description: Number of patients who undergo urgent/emergent surgical intervention post procedure
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cardioband
Number analyzed (Participants) | 11
Participants | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Cardioband
All-Cause Mortality (participants affected / at risk) | 5/11
Serious Adverse Events (participants affected / at risk) | 9/11
Other Adverse Events (participants affected / at risk) | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cardioband (N=11)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) — One patient experienced two Atrial Fibrillation adverse events (one serious and one non-serious). Both episodes are reported for this patient, one under Serious Adverse Events and the other under Other (Not Including Serious) Adverse Events.
Cardiac Failure (Cardiac disorders) | 6 (11)
Cardiac Failure Acute (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Large Intestine Polyp (Gastrointestinal disorders) | 1 (1)
Mechanical Ileus (Gastrointestinal disorders) | 1 (1)
General Physical Health Deterioration (General disorders) | 1 (1)
Bacterial Infection (Infections and infestations) | 1 (1)
Dermohypodermitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
IIIrd Nerve Disorder (Nervous system disorders) | 1 (1)
Device Malfunction (Product Issues) | 1 (1)
Completed Suicide (Psychiatric disorders) | 1 (1)
Haemorrhage Urinary Tract (Renal and urinary disorders) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Cervix Oedema (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Circulatory Collapse (Vascular disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Metabolic Disorder (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cardioband (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Heparin Induced Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (2) — One patient experienced two Atrial Fibrillation adverse events (one serious and one non-serious). Both episodes are reported for this patient, one under Serious Adverse Events and the other under Other (Not Including Serious) Adverse Events.
Supraventricular Tachycardia (Cardiac disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Creactive Protein Increased (Investigations) | 1 (1)
Haemoglobin Decreased (Investigations) | 2 (2)
Weight Increased (Investigations) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Puncture Site Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Tooth Infection (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 4 (4)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Depressed Level of Conciousness (Nervous system disorders) | 1 (1)
Device Pacing Issue (Product Issues) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypochromic Anaemia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/11/NCT02703311/Prot_SAP_000.pdf